CLINICAL TRIAL: NCT03080298
Title: International, Multicenter, Double-blind, Randomized, Placebo-controlled Phase 2a Study of the Efficacy and Safety of BP101 in Female Patients With Decrease or Loss of Sexual Desire
Brief Title: Study of the Efficacy and Safety of BP101 in Female Patients With Decrease or Loss of Sexual Desire
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ivix LLX (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP101-SD01
Record Dates: First submitted 2017-03-03; First posted 2017-03-15 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Hypoactive Sexual Desire Disorder (HSDD)
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with BP101 (Experimental)
  Interventions: Drug: BP101
- Treatment with placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BP101
  Arms: Treatment with BP101
Drug: Placebo
  Arms: Treatment with placebo

SUMMARY:
This is study of the efficacy, safety and pharmacokinetics of BP101 compared to placebo in patients with a decrease or loss of sexual desire.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 21 or older, who have signed informed concent, with a regular menstrual cycle (STRAW stages -5 to -3 (see Annex 7)).
* The level of follicle-stimulating hormone (FSH) is not more than 25 milli-International unit per ml (mIU/ml) according to the screening values.
* Decrease or loss of sexual desire (ICD-10 code: F-52.0) corresponding to the hypoactive sexual desire disorder (HSDD) diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM4), criteria.
* Current HSDD episode lasting not less than 24 weeks.
* Patients with secondary female sexual arousal disorder (FSAD) and/or female orgasmic disorder (FOD) will be eligible only if the HSDD developed before the FSAD and/or FOD and the HSDD has a more significant impact on the patient's quality of life.
* Not less than 15 scores according to the FSDS-R (Distress) Total Score.
* Stable monogamous relationship with one sexually active male sexual partner lasting at least a year. The partner is physically available not less than 50% of time during a month.
* Consent to attempt to have a sexual intercourse at least twice a month, if she has a desire.
* Consent to complete a diary every day during the screening period and assessment of the baseline state (in this period diary records must cover ≥80% days), during the therapy and subsequent follow-up.
* Consent to use adequate methods of contraception throughout the study.

Exclusion Criteria:

* Any prohibited treatments.
* Other mental disorders or psychiatric diseases.
* Score ≥ 20 according to the Beck Depression Inventory during the screening. Patients with 16 to 19 scores according to Beck's inventory may be included in the study unless, in the investigator's opinion, an actual depressive disorder is observed in the patient.
* Inflammatory diseases of pelvic organs, infections of the genitourinary system, cervicitis, interstitial cystitis, vulvodynia or severe atrophy of the vaginal epithelium.
* Surgical interventions (other than cosmetic surgeries) on reproductive organs in past medical history (ovariectomy, hysterectomy, obvious scars from childbirth-related perineal stitches, etc).
* Pregnant and nursing women or non-lactating women during the first 12 months after childbirth.
* Consumption of more than 5 portions of alcoholic drinks per week or alcohol addiction, drug addiction or drug abuse in the past. One portion of an alcoholic drink means 360 ml of beer, 120 ml of wine or 30 ml of a strong alcoholic drink.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Enrollment: 119 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
Desire domain score in the Female Sexual Function Index | 28 days (4 weeks) of treatment
  Change in the Desire domain score in the Female Sexual Function Index (FSFI) after 28 days (4 weeks) of treatment compared with the baseline.
Item 13 score in the Female Sexual Distress Scale-Revised | 28 days (4 weeks) of treatment
  Change of Item 13 score in the Female Sexual Distress Scale-Revised (FSDS-R) after 28 days (4 weeks) of treatment compared with the baseline.

SECONDARY OUTCOMES:
Desire domain in the Female Sexual Function Index | 28 days (4 weeks) of treatment and 56 days (8 weeks) of follow-up
  Change of the Desire domain in the Female Sexual Function Index (FSFI) after 28 days (4 weeks) and 56 days (8 weeks) of follow-up compared with the baseline.
Item 13 score in the Female Sexual Distress Scale-Revised | 28 days (4 weeks) of treatment and 56 days (8 weeks) of follow-up
  Change of Item 13 score in the Female Sexual Distress Scale-Revised (FSDS-R) after 28 days (4 weeks) and 56 days (8 weeks) of follow-up compared with the baseline.
Satisfying sexual events | 28 days (4 weeks) of treatment and 56 days (8 weeks) of follow-up
  Change in the number of satisfying sexual events (SSEs) in proportion to the 28 day period after 28 days (4 weeks) of the therapy and after 28 days (4 weeks) and 56 days (8 weeks) of follow-up compared with the baseline.
The total score of the Female Sexual Function Index | 28 days (4 weeks) of treatment and 56 days (8 weeks) of follow-up
  Change of the total score of the Female Sexual Function Index (FSFI) after 28 days (4 weeks) of the therapy and after 28 days (4 weeks) and 56 days (8 weeks) of follow-up compared with the baseline.
The total score of the Female Sexual Distress Scale-Revised | 28 days (4 weeks) of treatment and 56 days (8 weeks) of follow-up
  Change of total score of the Female Sexual Distress Scale-Revised (FSDS-R) after 28 days (4 weeks) of the therapy and after 28 days (4 weeks) and 56 days (8 weeks) of follow-up compared with the baseline.
The sexual function according to the Female Sexual Function questionnaire | 28 days (4 weeks) of treatment and 56 days (8 weeks) of follow-up
  Change of the sexual function according to the Female Sexual Function questionnaire (FSF) after 28 days (4 weeks) of the therapy and after 28 days (4 weeks) and 56 days (8 weeks) of follow-up compared with the baseline.
The patient's assessment of efficacy of the therapy according to the Patient Global Impression of Improvement | 28 days (4 weeks) of treatment and 56 days (8 weeks) of follow-up
  The patient's assessment of efficacy of the therapy according to the Patient Global Impression of Improvement (PGI-I) after 28 days (4 weeks) of the therapy and after 28 days (4 weeks) and 56 days (8 weeks) of the follow-up.
Number of adverse events | 28 days (4 weeks) of treatment and 56 days (8 weeks) of follow-up
  Frequency of adverse events reporting, including serious adverse events, in treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Daniil G Nemenov, MD, Study Director — IVIX Ltd.
Locations (12):
- Russia (12):
  - V.M. Bekhterev Republic Clinical Psychiatric Hospital, Kazan'
  - "People's Friendship University of Russia", Moscow
  - Mental Health Research Center, Moscow
  - N.A. Alexeev Moscow Psychiatric Clinical Hospital #1, Moscow
  - Clinical Psychiatry Hospital №1, Nizhny Novgorod
  - Orenburg Regional Clinical Psychiatric Hospital #1, Orenburg
  - OrKli Hospital LLC, Saint Petersburg
  - Regional Clinical Psychiatric Hospital of St. Sofia, Saratov
  - Engels Psycyatric hospital, Saratov Oblast
  - Clinic "Hundred Years", Tomsk
  - Yaroslavl Regional Clinical Psychiatric Hospital, Yaroslavl
  - Sverdlovsk Regional Clinical Psychiatric Hospital, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No